CLINICAL TRIAL: NCT02569385
Title: Examination of Cardiovascular Function/ Cardio Respiratory Interaction on Spontaneous Breathing Trials in Patients in the Prolonged Weaning
Acronym: Weaning TTE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: RWTH Aachen University (Other)
Responsible Party: Sponsor
Other Study IDs: CTC-A 15-034
Record Dates: First submitted 2015-09-23; First posted 2015-10-06 (Estimated); Last update posted 2015-10-06 (Estimated); Status verified 2015-08

CONDITIONS: Cardiovascular Disease
Keywords: Weaning TTE; patients in prolonged weaning
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- spontaneous breathing trials: spontaneous breathing trials in patients with prolonged weaning
  Interventions: Other: Spontaneous breathing trial

INTERVENTIONS:
Other: Spontaneous breathing trial

SUMMARY:
The aim of the present study is to determine the cardiovascular function/ cardio respiratory interaction on spontaneous breathing trials in patients with prolonged weaning.

ELIGIBILITY:
Inclusion Criteria:

* legal Age (≥18 years)
* written informed consent Prior to study participation
* patient in prolonged weaning with NYHA I-II and an actual positive Ventilator Screening test:

  1. PaO2 ≥ 60 mmHg at FiO2 ≤ 0.4
  2. PEEP ≤ 8 cmH2O
  3. Glasgow Coma Scale > 13
  4. Temp. < 38°C
  5. Hb > 80-100 g/L
  6. less requirement on catecholamines (<0.1µg/kg/min)
* and on these patients are already performed a spontaneous breathing trial with following result:

  1. abortion this spontaneous breathing trial < 30min, but possible > 10min
  2. reason for an abortion was NOT hypercapnia

Exclusion Criteria:

* weaning patients are assigned on Group 1-2
* patient with heart failure (NYHA III-IV) and/ or other cardiac comorbidity
* acute NSTEMI (non-ST-segment elevation myocardial infarction)
* pregnancy and breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients in prolonged weaning (Group 3 by Boles) with NYHA I-II, who come to the Department of Intensive Care Medicine RTWH Aachen University, will be recruited in the study. Recruitment will be performed in accordance to the inculsion and exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2015-08; Primary Completion 2016-08 (Estimated); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
Baseline measurement (Modus "CPAP-PS") in patient with prolonged weaning | 12 months
  under pressure support Ventilation are determined some measurement (e.g. breathing rate)

SECONDARY OUTCOMES:
Intervention measurement in patient with prolonged weaning | 12 months
  20 min breathing without mechanical ventilation

CONTACTS AND LOCATIONS:
Overall Officials: Michael Dreher, MD, Principal Investigator — Uniklinik RWTH Aachen, Med. Klinik I
Locations (1):
- University Hospital RWTH Aachen, Department of Medical Clinic I, Aachen, Germany